CLINICAL TRIAL: NCT02210169
Title: A Randomised Controlled Trial (RCT) of Continuous and Intermittent Infusion of Vancomycin in Neonates
Brief Title: RCT of Continuous Versus Intermittent Infusion of Vancomycin in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other); Royal Hospital For Women (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vanc_IIV vs CIV
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Sepsis; Infection; Bacteremia
MeSH Terms: conditions — Sepsis; Infections; Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent infusion of vancomycin (No Intervention): Vancomycin will be administered intravenously over 1 hour. Doses will be given from one to four times a day according to corrected gestational age.
- Continuous infusion of vancomycin (Active Comparator): A loading dose of vancomycin will be given over 1 hour followed by a continuous infusion of vancomycin over a 24 hour period.
  Interventions: Drug: Continuous infusion of vancomycin

INTERVENTIONS:
Drug: Continuous infusion of vancomycin — Continuous infusion of vancomycin will be given as a loading dose over 1 hour then as a continuous infusion over a 24-hours period.
  Arms: Continuous infusion of vancomycin

SUMMARY:
Babies aged 0 to 90 days with a suspected infection requiring treatment with vancomycin will be recruited. They will be randomised to receive vancomycin as an intermittent infusion (over 1 hour) or as a continuous infusion (over 24 hours). The hypothesis is that administering vancomycin as a continuous infusion will result in improved attainment of target concentrations in blood at steady state (when the drug is in equilibrium) compared to intermittent infusion.

ELIGIBILITY:
Inclusion Criteria:

- Neonates in the neonatal unit with an infection requiring treatment with vancomycin as determined by the treating physician.

Exclusion Criteria:

* Infants with a corrected gestational age < 25 weeks.
* Allergy to vancomycin or other glycopeptide antibiotic
* Vancomycin administered within the previous 72 hours
* Renal impairment
* Prior enrolment in the study
* Need for drug that is incompatible with vancomycin (if no other IV line is available)

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2014-09; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Proportion of neonates achieving target vancomycin concentrations in blood at steady state (24-48 hours) | 2 years

SECONDARY OUTCOMES:
Drug-related adverse effects | 2 years
  the proportion of drug-related adverse effects with CIV compared to IIV
Time to achieve target levels | 2 years
  the time to and number of dose adjustments required to achieve target therapeutic vancomycin levels in blood
Clearance of vancomycin in young infants | 2 years
  Population pharmacokinetic modelling of vancomycin in young infants using NONMEM
Volume of distribution of vancomycin in young infants | 2 years
  Population pharmacodynamics modelling of vancomycin in young infants using NONMEM
Area under the concentration-time curve of vancomycin in young infants | 2 years
  Population pharmacodynamics modelling of vancomycin in young infants using NONMEM
Time above the minimum inhibitory concentration of the bacteria for vancomycin in young infants | 2 years
  Population pharmacodynamics modelling of vancomycin in young infants using NONMEM

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Gwee, MBBS, Principal Investigator — Murdoch Childrens Research Institute
Locations (2):
- Australia (2):
  - Royal Hospital for Women, Sydney, New South Wales
  - The Royal Children's Hospital, Melbourne, Victoria

REFERENCES:
- [Derived] Gwee A, Cranswick N, McMullan B, Perkins E, Bolisetty S, Gardiner K, Daley A, Ward M, Chiletti R, Donath S, Hunt R, Curtis N. Continuous Versus Intermittent Vancomycin Infusions in Infants: A Randomized Controlled Trial. Pediatrics. 2019 Feb;143(2):e20182179. doi: 10.1542/peds.2018-2179. PMID 30700564
- [Derived] Gwee A, Cranswick N, Donath SM, Hunt R, Curtis N. Protocol for a randomised controlled trial of continuous infusions of vancomycin to improve the attainment of target vancomycin levels in young infants: The VANC trial. BMJ Open. 2018 Nov 3;8(11):e022603. doi: 10.1136/bmjopen-2018-022603. PMID 30391914